CLINICAL TRIAL: NCT03090295
Title: Does the Use of Both Palpation and Accuro as Compared to Palpation Alone or Use of Accuro Alone in a Single Patient Increase the First Pass Success Rate in Placing Spinals or Combined Spinal Epidurals for Cesarean Sections.
Brief Title: Palpation and ACCURO for Placing Spinal in C-section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Mohamed Tiouririne, MD, Associate Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 19713
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Anesthesia,Obstetrical
MeSH Terms: interventions — Palpation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Palpation and Accuro (Experimental): The placement site for the spinal anesthesia will be identified using both palpation and Accuro.
  Interventions: Device: Palpation and Accuro

INTERVENTIONS:
Device: Palpation and Accuro — Identify placement for spinal

SUMMARY:
The Accuro is a three dimensional handheld ultrasound device. This device uses sound waves to create pictures of the spine in three dimensions. This may allow the physician to view the spine in more detail for procedures such as spinal anesthesia and other diagnostic procedures.

We aim to assess the benefit of using both the Accuro and traditional landmark palpation technique to determine accurate spinal level in women who undergo cesarean section. This study will also assess provider preference for use of both Accuro and palpation compared with palpation alone or use of Accuro alone.

Anesthesia Providers will first identify the L4/L5 space using the traditional technique of palpating the iliac crests to estimate spinal level, which will be marked with a single dot from a marking pen. The provider will then use the Accuro 3000 to identify the L4/L5 interspace.

Results will be compared to results obtained in IRB 18070 "Handheld 3D lumbar spine navigation: A clinical validation study RM002" where subjects who were undergoing a C-section were randomized to either palpation or Accuro alone.

ELIGIBILITY:
Inclusion Criteria:

* • Patients between the ages of 18 and 45 presenting for a C-section delivery or scheduled for elective Cesarean section

  * ASA-1, ASA-2, and ASA-3
  * Patients with no known back deformities
  * Ability to sit upright for spinal placement
  * No prior lumbar surgery
  * No allergies to ultrasound gel

Exclusion Criteria:

* • Unable or unwilling to give informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
success rates | Day 1
  Success rates: defined as successful spinal administration on the first needle insertion attempt.

SECONDARY OUTCOMES:
Level of spinal placement: a record of the vertebral level where the spinal is administered. | Day 1
  Level of spinal placement: a record of the vertebral level where the spinal is administered.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Tiouririne, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chin KJ, Perlas A, Chan V, Brown-Shreves D, Koshkin A, Vaishnav V. Ultrasound imaging facilitates spinal anesthesia in adults with difficult surface anatomic landmarks. Anesthesiology. 2011 Jul;115(1):94-101. doi: 10.1097/ALN.0b013e31821a8ad4. PMID 21572316
- [Background] Vallejo MC, Phelps AL, Singh S, Orebaugh SL, Sah N. Ultrasound decreases the failed labor epidural rate in resident trainees. Int J Obstet Anesth. 2010 Oct;19(4):373-8. doi: 10.1016/j.ijoa.2010.04.002. Epub 2010 Aug 8. PMID 20696564
- [Background] Grau T, Leipold RW, Conradi R, Martin E. Ultrasound control for presumed difficult epidural puncture. Acta Anaesthesiol Scand. 2001 Jul;45(6):766-71. doi: 10.1034/j.1399-6576.2001.045006766.x. PMID 11421838
- [Background] Grau T, Bartusseck E, Conradi R, Martin E, Motsch J. Ultrasound imaging improves learning curves in obstetric epidural anesthesia: a preliminary study. Can J Anaesth. 2003 Dec;50(10):1047-50. doi: 10.1007/BF03018371. PMID 14656785
- [Background] Chin KJ, Karmakar MK, Peng P. Ultrasonography of the adult thoracic and lumbar spine for central neuraxial blockade. Anesthesiology. 2011 Jun;114(6):1459-85. doi: 10.1097/ALN.0b013e318210f9f8. PMID 21422997
- [Background] Karmakar MK. Ultrasound for central neuroaxial blocks. Techniques in regional anesthesia and pain management 2009;13:161-70.